CLINICAL TRIAL: NCT01873248
Title: Impact of 68Ga-DOTATATE PET/CT on the Management of Neuroendocrine Tumors: The Referring Physician's Perspective
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-001920; 68Ga-DOTATATE PET/CT (Other: Jonsson Comprehensive Cancer Center); NCI-2016-01796 (Registry Identifier: CTRP)
Expanded Access: NCT02174679 (No longer available)
Record Dates: First submitted 2013-06-03; First posted 2013-06-10 (Estimated); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Neuroendocrine Tumors
Keywords: NET; neuroendocrine tumors; somastostatin receptor; PET; DOTATATE
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET/CT with one-time administration of 68Ga-DOTATATE (Experimental): Study participants will receive a one-time administration of 68Ga-DOTATATE and undergo a PET/CT imaging study. Scans will be performed with oral and IV contrast. The physicians of patient's receiving a 68Ga-DOTATATE PET/CT will be asked to fill out 2 questionnaires with questions pertaining to the patient's medical management. One questionnaire will be sent before the scan, and one shortly after the scan was performed and the results reported to the referring physician.
  Interventions: Drug: 68Ga-DOTATATE

INTERVENTIONS:
Drug: 68Ga-DOTATATE — 68Ga-DOTATATE will be given in tracer doses and injected intravenously to image Neuroendocrine tumors by Positron Emission Tomography.
  Other Names: 68Ga-DOTATATE PET/CT scan

SUMMARY:
Somatostatin receptor imaging with 68Ga-DOTATATE PET/CT (DOTATATE) is increasingly used for managing patients with neuroendocrine tumors. The objective of this study was to determine referring physicians' perspectives on the impact of DOTATATE on the management of neuroendocrine tumors.

DETAILED DESCRIPTION:
Somatostatin receptor imaging with 68Ga-DOTATATE PET/CT (DOTATATE) is increasingly used for managing patients with neuroendocrine tumors. The objective of this study was to determine referring physicians' perspectives on the impact of DOTATATE on the management of neuroendocrine tumors. Methods: A set of 2 questionnaires (pre-PET and post-PET) was sent to the referring physicians of 100 consecutive patients with known or suspected neuroendocrine tumors, who were evaluated with DOTATATE. Questionnaires on 88 patients were returned (response rate, 88%). Referring physicians categorized the DOTATATE findings on the basis of the written PET reports as negative, positive, or equivocal for disease. The likelihood for metastatic disease was scored as low, moderate, or high. The intended management before and changes as a consequence of the PET study were indicated. Results: The indications for PET/CT were initial and subsequent treatment strategy assessments in 14% and 86% of patients, respectively. Referring physicians reported that DOTATATE led to a change in suspicion for metastatic disease in 21 patients (24%; increased and decreased suspicion in 9 [10%] and 12 [14%] patients, respectively). Intended management changes were reported in 53 of 88 (60%) patients. Twenty patients (23%) scheduled to undergo chemotherapy were switched to treatments without chemotherapy, and 6 (7%) were switched from watch-and-wait to other treatment strategies. Conversely, 5 patients (6%) were switched from their initial treatment strategy to watch-and-wait. Conclusion: This survey of referring physicians demonstrates a substantial impact of DOTATATE on the intended management of patients with neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of NET, suspected SSTR positive tumors or suspected NET recurrence.
* At least 18 years of age.
* Patient or patient's legally acceptable representative cognitively provides written informed consent.
* Able to provide informed consent.
* Females of childbearing potential must have a negative pregnancy test at screening/baseline.

Exclusion Criteria:

* Use of any other investigational product or device within 30 days prior to dosing, or known requirement for any other investigational agent prior to completion of all scheduled study assessments.
* Patients with a body weight of 400 pounds or more or not able to enter the bore of the PET/CT scanner due to BMI, because of the compromise in image quality with CT, PET/CT and MRI that will result.
* Inability to lie still for the entire imaging time.
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Recognized concurrent active infection.
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08-26 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Change in intended management of patients with NETs after PET/CT | Before the first scan and after the second scan and results reported
  The study will collect questionnaire data from referring physicians on intended patient management before and after PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Nuclear Medicine Clinic of the Department of Molecular and Medical Pharmacology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modlin IM, Moss SF, Chung DC, Jensen RT, Snyderwine E. Priorities for improving the management of gastroenteropancreatic neuroendocrine tumors. J Natl Cancer Inst. 2008 Sep 17;100(18):1282-9. doi: 10.1093/jnci/djn275. Epub 2008 Sep 9. PMID 18780869
- [Background] Modlin IM, Oberg K, Chung DC, Jensen RT, de Herder WW, Thakker RV, Caplin M, Delle Fave G, Kaltsas GA, Krenning EP, Moss SF, Nilsson O, Rindi G, Salazar R, Ruszniewski P, Sundin A. Gastroenteropancreatic neuroendocrine tumours. Lancet Oncol. 2008 Jan;9(1):61-72. doi: 10.1016/S1470-2045(07)70410-2. PMID 18177818
- [Background] Yao JC, Hassan M, Phan A, Dagohoy C, Leary C, Mares JE, Abdalla EK, Fleming JB, Vauthey JN, Rashid A, Evans DB. One hundred years after "carcinoid": epidemiology of and prognostic factors for neuroendocrine tumors in 35,825 cases in the United States. J Clin Oncol. 2008 Jun 20;26(18):3063-72. doi: 10.1200/JCO.2007.15.4377. PMID 18565894
- [Background] Rensing BJ, Hermans WR, Strauss BH, Serruys PW. Regional differences in elastic recoil after percutaneous transluminal coronary angioplasty: a quantitative angiographic study. J Am Coll Cardiol. 1991 May;17(6 Suppl B):34B-38B. doi: 10.1016/0735-1097(91)90936-4. PMID 2016480
- [Background] Virgolini I, Ambrosini V, Bomanji JB, Baum RP, Fanti S, Gabriel M, Papathanasiou ND, Pepe G, Oyen W, De Cristoforo C, Chiti A. Procedure guidelines for PET/CT tumour imaging with 68Ga-DOTA-conjugated peptides: 68Ga-DOTA-TOC, 68Ga-DOTA-NOC, 68Ga-DOTA-TATE. Eur J Nucl Med Mol Imaging. 2010 Oct;37(10):2004-10. doi: 10.1007/s00259-010-1512-3. PMID 20596866
- [Background] Kowalski J, Henze M, Schuhmacher J, Macke HR, Hofmann M, Haberkorn U. Evaluation of positron emission tomography imaging using [68Ga]-DOTA-D Phe(1)-Tyr(3)-Octreotide in comparison to [111In]-DTPAOC SPECT. First results in patients with neuroendocrine tumors. Mol Imaging Biol. 2003 Jan-Feb;5(1):42-8. doi: 10.1016/s1536-1632(03)00038-6. PMID 14499161
- [Background] Hofmann M, Maecke H, Borner R, Weckesser E, Schoffski P, Oei L, Schumacher J, Henze M, Heppeler A, Meyer J, Knapp H. Biokinetics and imaging with the somatostatin receptor PET radioligand (68)Ga-DOTATOC: preliminary data. Eur J Nucl Med. 2001 Dec;28(12):1751-7. doi: 10.1007/s002590100639. Epub 2001 Oct 31. PMID 11734911
- [Background] Gabriel M, Decristoforo C, Kendler D, Dobrozemsky G, Heute D, Uprimny C, Kovacs P, Von Guggenberg E, Bale R, Virgolini IJ. 68Ga-DOTA-Tyr3-octreotide PET in neuroendocrine tumors: comparison with somatostatin receptor scintigraphy and CT. J Nucl Med. 2007 Apr;48(4):508-18. doi: 10.2967/jnumed.106.035667. PMID 17401086
- [Background] Putzer D, Gabriel M, Henninger B, Kendler D, Uprimny C, Dobrozemsky G, Decristoforo C, Bale RJ, Jaschke W, Virgolini IJ. Bone metastases in patients with neuroendocrine tumor: 68Ga-DOTA-Tyr3-octreotide PET in comparison to CT and bone scintigraphy. J Nucl Med. 2009 Aug;50(8):1214-21. doi: 10.2967/jnumed.108.060236. Epub 2009 Jul 17. PMID 19617343
- [Background] Prasad V, Ambrosini V, Hommann M, Hoersch D, Fanti S, Baum RP. Detection of unknown primary neuroendocrine tumours (CUP-NET) using (68)Ga-DOTA-NOC receptor PET/CT. Eur J Nucl Med Mol Imaging. 2010 Jan;37(1):67-77. doi: 10.1007/s00259-009-1205-y. PMID 19618183
- [Background] Ambrosini V, Tomassetti P, Franchi R, Fanti S. Imaging of NETs with PET radiopharmaceuticals. Q J Nucl Med Mol Imaging. 2010 Feb;54(1):16-23. PMID 20168283
- See also: Ahmanson Imaging Division — http://www.pet.ucla.edu
- See also: Department of Molecular and Medical Pharmacology UCLA — http://www.pharmacology.ucla.edu